CLINICAL TRIAL: NCT01347697
Title: Nordic Extended Abdominoperineal Excision (NEAPE) Study, a RCT Comparing a Porcine Acellular Dermal Collagen Implant (Biological Mesh) With a Gluteus Maximus Flap for Reconstruction of Pelvic Floor After ELAPE in Rectal Cancer
Brief Title: Collagen Implant (Biological Mesh) Versus GM Flap for Reconstruction of Pelvic Floor After ELAPE in Rectal Cancer
Acronym: NEAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: The Swedish Society of Medicine (Other); Västerbotten County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEAPE-2010-335-31M
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer; Defect of Floor of Lesser Pelvis
Keywords: rectal neoplasms; reconstructive surgical procedure; bioprosthesis; surgical flaps; locomotion; lesser pelvis
MeSH Terms: conditions — Rectal Neoplasms | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Porcine collagen implant (biological mesh) (Experimental): Reconstruction with an acellular porcine dermal collagen implant (biological mesh).
  Interventions: Procedure: Reconstruction with an acellular porcine dermal collagen implant (biological mesh)
- Gluteus maximus flap (Active Comparator): Reconstruction with a gluteus maximus myocutaneous flap.
  Interventions: Procedure: Reconstruction with a gluteus maximus myocutaneous flap

INTERVENTIONS:
Procedure: Reconstruction with an acellular porcine dermal collagen implant (biological mesh) — Reconstruction of floor of lesser pelvis with an acellular porcine dermal collagen implant (biological mesh) after extended excision of rectum including levator muscles in advanced low rectal cancer.
  Arms: Porcine collagen implant (biological mesh)
Procedure: Reconstruction with a gluteus maximus myocutaneous flap — Reconstruction of floor of lesser pelvis with an gluteus maximus myocutaneous flap after extended excision of rectum including levator muscles in advanced low rectal cancer.
  Arms: Gluteus maximus flap

SUMMARY:
The trial compares two different techniques for reconstruction of the lesser pelvic floor after an extended abdominoperineal excision for locally advanced rectal cancer. The alternative reconstruction techniques in the trial are:

* a technique using a gluteus maximus myocutaneous flap or
* a technique using an acellular porcine collagen implant (biological mesh)

The primary endpoint will be physical performance six months from operation and our hypothesis is that the technique using an acellular porcine implant will cause less impaired physical performance compared to the technique using a myocutaneous flap.

The study is interventional, randomized and by definition a comparative effectiveness research project.

DETAILED DESCRIPTION:
Extended abdominoperineal excision (EAPE) of the rectum is the potentially curative operation for rectal carcinomas too low for primary anastomosis, especially if the levator and sphincter musculature is infiltrated. This enlarged operation, when the levator musculature is excised en bloc with the rectum, creates a large defect. Primary closure is often not possible, and reconstruction with prosthetic material or a myocutaneous flap is necessary to avoid a perineal hernia. Implantation of a collagen sheet (biological mesh) has shown preliminary good results and on the other hand, the use of a gluteus myocutaneous flap is routine in many clinics. There is a lack of scientific evidence to prove which method is better for the reconstruction of the lesser pelvic floor.

The current study aims to compare the two reconstruction techniques.

Centres that treat locally advanced rectal cancers with the extended abdominoperineal excision of rectum (EAPE)[Holm et al 2007] can participate provided that:

1. the operative technique is standardized according to the study protocol
2. the centre/unit has resources for examinations of participants by a physiotherapist or a nurse
3. the centre/unit has one investigator in charge of the study locally
4. the centre/unit has an operative volume that enables at least 6 patients to be included/randomised during the anticipated three year study phase for inclusions

Centres that do not operate the rectal cancers included in this study can participate by arranging the preoperative examination and physical tests as well as follow-up of patients that are referred to other centres for the operation. In these cases the operating centre cares for the randomisation, operation and start of postoperative rehabilitation while the study follow-up and final rehabilitation can be completed at the patients' primary referral hospital. The primary referral hospital needs a site investigator in charge of study patients just like centres that do the operations.

Patients with primary or recurrent cancers of rectal origin can be included but individual patients can be included only once. Concomitant therapies are allowed and preoperative or postoperative radiation therapy and/or chemotherapy may be given or not according to local multidisciplinary team (MDT) decisions.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) rectal cancer patients where wide resection of pelvic floor muscles together with rectum and anal canal have made reconstruction of pelvic floor necessary i.e. primary suture of pelvic floor in the midline is not possible. Resection of coccyx is optional.

Exclusion Criteria:

* Age less than 18 years
* Very large resections including partial resection of sacrum and patients considered for bilateral flap reconstruction
* Large concomitant resection of vaginal wall where total (vaginal) wound closure is not an option
* Expected survival less than one year at operation
* Patient do not sign informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Performance in Timed-Stands Test | 6 months after surgery
  Timed-Stands test is a combined measure of physical performance depending on at least muscle strength, balance, tenderness of gluteal skin and muscles and co-ordination of motion.

SECONDARY OUTCOMES:
Change in physical performance | 3, 6 and 12 months after surgery compared with preoperative results
  Change in Timed-Stands Test performance
Primary wound healing assessed with the Southampton Wound Assessment Scale | 3 months from operation
  The Southampton Wound Assessment Scale is a validated measure of wound healing after surgery.
Complications according to classification by Dindo-Clavien | 3, 6 and 12 months after surgery
  The Dindo-Clavien classification of surgical complications is a validated instrument.
Proportion of persistent perineal sinus or fistula | 3, 6 and 12 months after surgery
  Proportion of patients with the wound healing defect of all patients in the particular study arm
Ability to sit | 3, 6 and 12 months after surgery
  Ability to sit is graded with a scale in three degrees.
Change of pain and discomfort in gluteal region measured with VAS | 3, 6 and 12 months after surgery compared to preoperative
  A standard visual analogue scale (VAS) from 0-100 mm is used.
Pain and discomfort in gluteal region, spot measures with VAS | 3, 6 and 12 months after surgery
  A standard visual analogue scale (VAS) from 0-100 mm is used.
Change of quality of life measured with EQ-5D and EORTC forms C30 and CR29 | 3, 6 and 12 months after surgery compared to preoperative
  EQ-5D and EORTC are validated quality of life instruments
Quality of life spot measures | 3, 6 and 12 months after surgery
  Quality of life at specified time points
Length of hospital stay | Six months after surgery
  Length of index hospital stay in days.
Costs of surgical treatment | 12 months after surgery
  Hospital expenses converted to US$
Quality-adjusted life years (QALYs gained) | 12 months after surgery
  Quality adjusted life year (QALY) is calculated using an quality of life utility index at repeated time points. The utility index is adjusted for the relevant background population.
Local recurrence | Five years after surgery
  Local recurrence of rectal cancer detected by clinical or radiological investigation

CONTACTS AND LOCATIONS:
Overall Officials: Markku M Haapamäki, MD, PhD, Principal Investigator — Umeå University, Department of Surgical and Perioperative Sciences; Jörgen Rutegård, MD, PhD, Study Director — Umeå University
Locations (8):
- Oulu University Hospital, Oulu, Finland
- Sweden (7):
  - Sunderby County Hospital, Luleå
  - Skåne Universtiy Hospital, Malmo
  - Östersund Hospital, Östersund
  - Karolinska University Hospital, Solna, Stockholm
  - Umeå University Hospital, Department of Surgical and Perioperative Sciences, Umeå
  - Uppsala University Hospital, Uppsala
  - Västmanlands Sjukhus Västerås, Västerås

REFERENCES:
- [Background] Holm T, Ljung A, Haggmark T, Jurell G, Lagergren J. Extended abdominoperineal resection with gluteus maximus flap reconstruction of the pelvic floor for rectal cancer. Br J Surg. 2007 Feb;94(2):232-8. doi: 10.1002/bjs.5489. PMID 17143848
- [Background] Haapamaki MM, Pihlgren V, Lundberg O, Sandzen B, Rutegard J. Physical performance and quality of life after extended abdominoperineal excision of rectum and reconstruction of the pelvic floor with gluteus maximus flap. Dis Colon Rectum. 2011 Jan;54(1):101-6. doi: 10.1007/DCR.0b013e3181fce26e. PMID 21160320
- [Derived] Rutegard M, Rutegard J, Haapamaki MM. Multicentre, randomised trial comparing acellular porcine collagen implant versus gluteus maximus myocutaneous flap for reconstruction of the pelvic floor after extended abdominoperineal excision of rectum: study protocol for the Nordic Extended Abdominoperineal Excision (NEAPE) study. BMJ Open. 2019 May 29;9(5):e027255. doi: 10.1136/bmjopen-2018-027255. PMID 31147361